CLINICAL TRIAL: NCT01612858
Title: Metabolic Abnormalities in HIV-infected Persons
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLAMP-K23; 1K23DK079789-01A2 (NIH)
Record Dates: First submitted 2012-06-04; First posted 2012-06-06 (Estimated); Results first posted 2016-06-20 (Estimated); Last update posted 2016-06-20 (Estimated); Status verified 2016-05

CONDITIONS: Lipodystrophy; HIV Infection
Keywords: Lipodystrophy; Insulin resistance; HIV infection
MeSH Terms: conditions — Lipodystrophy; HIV Infections; Insulin Resistance | interventions — Metformin; Pioglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metformin (Experimental)
  Interventions: Drug: Metformin
- Pioglitazone (Experimental)
  Interventions: Drug: Pioglitazone

INTERVENTIONS:
Drug: Metformin — Metformin at a dose of one 500mg tablet twice a day with meals for one week, after which the dose will increase to 500 mg three times a day with meals for the remaining 11 weeks of the study.
  Other Names: Fortamet; Glucophage; Glumetza; Riomet
  Arms: Metformin
Drug: Pioglitazone — Pioglitazone at a dose of one 30 mg tablet once per day for the 12 weeks of the study.
  Other Names: Actos
  Arms: Pioglitazone

SUMMARY:
The purpose of this study is to examine the relationship between insulin resistance and changes in body fat distribution in HIV-infected persons. This study measures insulin sensitivity, abdominal fat, and intramuscular fat in HIV-infected persons and examines the effect of an anti-diabetic drug (metformin or pioglitazone) on insulin sensitivity and body fat in this population.

DETAILED DESCRIPTION:
Although HIV antiretroviral medications have helped patients live longer, they have also been associated with side effects including insulin resistance and changes in body fat distribution. Changes in body fat distribution associated with HIV antiretroviral medications may result in increased fat in the abdomen, neck, and upper back, which is often called central fat deposition. HIV antiretroviral medications may also result in loss of fat in legs, arms, and face, which is often called peripheral fat atrophy.

This study will obtain preliminary data on the effect of 12 weeks of metformin on insulin sensitivity and hepatic and peripheral muscle fat in HIV-infected persons with insulin resistance and central fat deposition. Similarly, this study will obtain preliminary data on the effect of 12 weeks of pioglitazone on insulin sensitivity and hepatic and peripheral muscle fat in HIV-infected persons with insulin resistance and peripheral fat atrophy.

This study involves taking a drug that has been approved by the U.S. Food and Drug Administration (FDA) for use in humans for a period of 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years
* Fasting insulin >12 μU/mL and/or serum glucose between 140-200 mg/dl after 75 g 2hr oral glucose tolerance test
* Central fat deposition or Peripheral fat atrophy
* Fasting glucose ≤126 mg/dL
* BMI ≥18 and ≤35 kg/m2
* CD4 cell count ≥100 cells/mm3
* Stable antiretroviral regimen ≥12 weeks and HIV RNA <1000 copies

Exclusion Criteria:

* Diabetes mellitus
* Cardiac pacemaker or metal implant
* Liver enzymes >2.5x upper normal limit
* Alkaline phosphatase or prothrombin time >2x upper normal limit
* Serum creatinine >1.4 mg/dL
* History of congestive heart failure
* Hemoglobin <8 g/dL
* Alcohol abuse
* Pregnancy
* History of lactic acidosis
* Use of steroids
* Acute infection within last one month
* History of bladder cancer

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-06; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rakhi Kohli, MD, MS, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Metformin | Pioglitazone
Started | 16 | 4
Completed | 11 | 3
Not Completed | 5 | 1
Not completed — Withdrawal by Subject | 5 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metformin | Pioglitazone | Total
Number analyzed (Participants) | 16 | 4 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.9 (7.9) | 55.7 (8.6) | 54.2 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 0 | 4
  Male | 12 | 4 | 16

OUTCOME MEASURES:

1. Primary Outcome: Change in Insulin Sensitivity From Baseline to Week 12 Post-treatment With Insulin Sensitizing Agent
Description: Change in insulin sensitivity measured by 2 hour euglycemic-hyperinsulinemic clamp from baseline to week 12 post treatment with metformin or pioglitazone
Time Frame: 3 months
Population: Only participants with baseline and post insulin-sensitizing treatment euglycemic-hyperinsulinemic clamp were included in this analysis
Measure: Mean (Standard Deviation); unit: mg/kg lean body mass/min
Arm/Group | Metformin | Pioglitazone
Number analyzed (Participants) | 11 | 3
mg/kg lean body mass/min | -0.25 (1.98) | -0.96 (0.43)

2. Secondary Outcome: Change in Hepatic Fat From Baseline to Week 12 Post-treatment With an Insulin Sensitizing Agent
Description: Change in hepatic fat was measured after 12 weeks of treatment with metformin or pioglitazone using magnetic resonance spectroscopy
Time Frame: 12 weeks
Population: Only participants with baseline and post insulin sensitizing treatment magnetic resonance spectrosocpy were included in this analysis.
Measure: Mean (Standard Deviation); unit: percentage of hepatic fat
Arm/Group | Metformin | Pioglitazone
Number analyzed (Participants) | 11 | 3
percentage of hepatic fat | 2.30 (2.10) | -2.56 (1.16)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for three months.
Arm/Group | Metformin | Pioglitazone
Serious Adverse Events (participants affected / at risk) | 7/16 | 0/4
Other Adverse Events (participants affected / at risk) | 4/16 | 1/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metformin (N=16) | Pioglitazone (N=4)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Elevated serum creatinine (Renal and urinary disorders) | 2 (2) | 0 — Two subjects experienced asymptomatic elevation in serum creatinine within 1.5 times the upper limit of normal.
Elevated lactic acid (Metabolism and nutrition disorders) | 2 (2) | 0 — Two subjects developed asymptomatic elevation in lactic acid between 1.5 and 2 times the upper limit of normal.
Right upper quadrant abdominal pain (Gastrointestinal disorders) | 1 (1) | 0
Head trauma accompanied by syncope (Nervous system disorders) | 1 (1) | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metformin (N=16) | Pioglitazone (N=4)
Bloating (Gastrointestinal disorders) | 1 (1) | 0
diarrhea (Gastrointestinal disorders) | 3 (3) | 1 (1)
vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Baker's cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0
tooth pain (Infections and infestations) | 1 (1) | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No